CLINICAL TRIAL: NCT06588647
Title: Efficacy of the Improving Participation After Stroke Self-Management-Rehabilitation (IPASS-R) Program in Sub-acute Stroke
Brief Title: Improving Participation After Stroke Self-Management-Rehabilitation
Acronym: IPASS-R
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: University of Washington (Other); National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Anna Boone, Assistant Professor of Occupational Therapy, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2108606; 1R01HD114732-01 (NIH)
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Stroke
Keywords: Stroke; Self-Management; Telehealth; Activities of daily living; Community engagement
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All outcomes assessors will be blinded to participant study group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Improving Participation after Stroke Self-Management Program (IPASS) (Experimental): The IPASS-R intervention consists of 6 weekly 90-minute sessions delivered by an occupational therapist and stroke survivor peer facilitator. All sessions will be delivered remotely via videoconferencing.
  Interventions: Behavioral: Improving Participation after Stroke Self-Management Program (IPASS)
- Chronic Disease Self-Management Program (CDSMP) (Active Comparator): The CDSMP will consist of 6, weekly 90-minute sessions. All sessions will be delivered remotely via videoconferencing.
  Interventions: Behavioral: Chronic Disease Self-Management Program (CDSMP)

INTERVENTIONS:
Behavioral: Improving Participation after Stroke Self-Management Program (IPASS) — The IPASS-R program is a group-based self-management intervention that aims to improve problem-solving, action-planning, and resource utilization skills for improved community living and participation. The Activity-Barriers-Changes-Doing-Evaluation (ABCDE) framework is a user friendly problem-solving and goal setting framework that is used repetitively in each session throughout the program. Participants are guided to identify (1) an activity that they want to improve or re-engage in (A); (2) individual and environmental barriers that hinder their engagement (B); (3) changes that they can make to deal with the barriers and improve their engagement (C); and (4) an action plan to pursue (D). After the action plan, participants come back in the next session and evaluate their performance in following through on their plans (E).
  Arms: Improving Participation after Stroke Self-Management Program (IPASS)
Behavioral: Chronic Disease Self-Management Program (CDSMP) — The program is facilitated by two trained leaders in small groups in a community setting with individuals who have chronic health problems and will follow the CDSMP protocol. Participants receive education on various health-related topics applicable to a range of chronic conditions, share experiences, and support one another.
  Arms: Chronic Disease Self-Management Program (CDSMP)

SUMMARY:
The overall goal of this proposed study is to evaluate the efficacy of a small-group, stroke-specific, self-management program delivered via telehealth to improve self-efficacy, activity performance, and quality of life in individuals with sub-acute stroke.

ELIGIBILITY:
Inclusion Criteria:

* less than 6 months post-stroke
* age 45-85 years
* completed inpatient rehabilitation services (if recommended)
* living in the community with or without caregiver support (i.e., not living in a skilled nursing facility)
* ability to read, write, and speak English
* diagnosis of mild or moderate stroke (National Institutes of Health stroke score <16)
* able to use videoconferencing independently or with caregiver support

Exclusion Criteria:

* severe depressive symptoms as indicated by a score ≥21 on the Patient Health Questionnaire
* dementia symptoms as indicated by a score of <23 on the Montreal Cognitive Assessment
* additional neurological diagnoses (e.g., brain malignancy, previous severe stroke)
* (4) moderate or severe aphasia as indicated by a National Institutes of Health Stroke Scale aphasia score of ≥ 2
* inability to provide informed consent
* any other condition not otherwise specified that the PI determines would render participation in this study as unsafe for the participant

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2029-12-15 (Estimated); Study Completion 2029-12-15 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) Performance | Pre-intervention (week 0), post-intervention (week 6), and 6-month follow-up (week 32)
  Self-report measure of activity performance. Minimum = 1, Maximum = 10. Higher scores mean better performance.
Canadian Occupational Performance Measure (COPM) Satisfaction | Pre-intervention (week 0), post-intervention (week 6), and 6-month follow-up (week 32)
  Self-report measure of activity performance. Minimum = 1, Maximum = 10. Higher scores mean higher satisfaction.
Participation Strategies Self-Efficacy Scale (PS-SES) | Pre-intervention (week 0), post-intervention (week 6), and 6-month follow-up (week 32)
  Self-report measure of self-efficacy in using participation strategies. The subject rates confidence across 35 items within six subscales: (1) managing home participation, (2) staying organized, (3) planning and managing community participation, (4) managing work and productivity), (5) managing communication, and (6) advocating for resources. Range of scores from 35-350. Higher scores indicate greater self-efficacy.

SECONDARY OUTCOMES:
In home activity level as measured by sensor system | Duration of study (from baseline assessment (week 0) to 6-month follow-up assessment)
  average hourly percentage of time spent engaged in activity
Community engagement as measured by sensor system | Duration of study (from baseline assessment (week 0) to 6-month follow-up assessment)
  Time outside the home as measured by time between door sensor activations
Stroke Impact Scale participation domain | Pre-intervention (week 0), post-intervention (week 6), and 6-month follow-up (week 32)
  Measures perceived stroke recovery/quality of life. Range of scores 0-100. Higher scores indicate higher performance.
Assessment of Life Habits (LIFE-H) | Pre-intervention (week 0), post-intervention (week 6), and 6-month follow-up (week 32)
  Measures self-reported participation in daily activities by measuring total score across 6 domains. Score range of 0 to 9 with higher scores indicating better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Anna E Boone, PhD, OTR/L, Principal Investigator — University of Missouri Occupational Therapy
Locations (1):
- University of Missouri, Columbia, Missouri, United States

REFERENCES:
- [Background] Jette DU, Latham NK, Smout RJ, Gassaway J, Slavin MD, Horn SD. Physical therapy interventions for patients with stroke in inpatient rehabilitation facilities. Phys Ther. 2005 Mar;85(3):238-48. PMID 15733048
- [Background] Sakakibara BM, Kim AJ, Eng JJ. A Systematic Review and Meta-Analysis on Self-Management for Improving Risk Factor Control in Stroke Patients. Int J Behav Med. 2017 Feb;24(1):42-53. doi: 10.1007/s12529-016-9582-7. PMID 27469998
- [Background] Fryer CE, Luker JA, McDonnell MN, Hillier SL. Self management programmes for quality of life in people with stroke. Cochrane Database Syst Rev. 2016 Aug 22;2016(8):CD010442. doi: 10.1002/14651858.CD010442.pub2. PMID 27545611
- [Background] Chen L, Chen Y, Chen X, Shen X, Wang Q, Sun C. Longitudinal Study of Effectiveness of a Patient-Centered Self-Management Empowerment Intervention During Predischarge Planning on Stroke Survivors. Worldviews Evid Based Nurs. 2018 Jun;15(3):197-205. doi: 10.1111/wvn.12295. PMID 29878691
- [Background] Cadilhac DA, Hoffmann S, Kilkenny M, Lindley R, Lalor E, Osborne RH, Batterbsy M. A phase II multicentered, single-blind, randomized, controlled trial of the stroke self-management program. Stroke. 2011 Jun;42(6):1673-9. doi: 10.1161/STROKEAHA.110.601997. Epub 2011 Apr 14. PMID 21493910
- [Background] Wolf TJ, Baum CM, Lee D, Hammel J. The Development of the Improving Participation after Stroke Self-Management Program (IPASS): An Exploratory Randomized Clinical Study. Top Stroke Rehabil. 2016 Aug;23(4):284-92. doi: 10.1080/10749357.2016.1155278. Epub 2016 Mar 16. PMID 27077987
- [Background] Lee D, Fischer H, Zera S, Robertson R, Hammel J. Examining a participation-focused stroke self-management intervention in a day rehabilitation setting: a quasi-experimental pilot study. Top Stroke Rehabil. 2017 Dec;24(8):601-607. doi: 10.1080/10749357.2017.1375222. Epub 2017 Sep 28. PMID 28956721